CLINICAL TRIAL: NCT00927225
Title: Local Infiltration Analgesia in Bilateral Knee Arthroplasty - Efficacy of Subcutaneous Wound Infiltration With Local Anesthetic.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Lasse Andersen, Hvidovre Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-D-2008-104
Record Dates: First submitted 2009-06-23; First posted 2009-06-24 (Estimated); Last update posted 2009-06-24 (Estimated); Status verified 2009-06

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- active (Active Comparator): subcutaneous wound infiltration with 50 mL ropivacaine 0.2%
  Interventions: Drug: ropivacaine 0.2%, 50 mL
- placebo (Placebo Comparator): subcutaneous wound infiltration with 50 mL saline
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: ropivacaine 0.2%, 50 mL
  Arms: active
Drug: normal saline
  Arms: placebo

SUMMARY:
Local infiltration analgesia is effective in total knee arthroplasty for postoperative pain management, but the efficacy of subcutaneous wound infiltration has not been evaluated. This study aims at evaluating the efficacy of subcutaneous wound infiltration in total knee arthroplasty in 16 patients undergoing bilateral knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* total bilateral knee arthroplasty

Exclusion Criteria:

* immunological diseases
* treatment with opioids or steroids
* allergy to any drugs administered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 1-6 hours postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

REFERENCES:
- [Derived] Andersen LO, Husted H, Kristensen BB, Otte KS, Gaarn-Larsen L, Kehlet H. Analgesic efficacy of subcutaneous local anaesthetic wound infiltration in bilateral knee arthroplasty: a randomised, placebo-controlled, double-blind trial. Acta Anaesthesiol Scand. 2010 May;54(5):543-8. doi: 10.1111/j.1399-6576.2009.02196.x. Epub 2010 Jan 6. PMID 20055763